CLINICAL TRIAL: NCT05388604
Title: Prospective Clinical Study To Evaluate The Efficacy And Safety Of Paired Treatment With A Picosecond 755nm Alexandrite Laser With Focused Lens Array And Radiofrequency Microneedling For Facial Aging
Brief Title: Clinical Study To Evaluate Paired Treatment With An Alexandrite Laser And Radiofrequency Microneedling For Facial Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD-PM01-2021
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Wrinkle; Photoaging; Dyschromia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Subjects are to be treated with the RF device, followed by the microneedling device. Parameters may be adjusted throughout the treatment and will determined by the Clinician. Subjects will receive up to 4 treatments, spaced approximately 4 weeks apart.
  Interventions: Device: RF device; Device: Microneedling device

INTERVENTIONS:
Device: RF device — The entire defined treatment area will then be treated by delivering adjacent pulses with minimal overlap of 10% or less. Parameters may be adjusted throughout the treatment in order to increase subject comfort.
Device: Microneedling device — Test spots may be performed prior to the first treatment. Test spots may be performed prior to the first treatment. It will follow a similar procedure to treatment but only in an inconspicuous place, such as behind the ear, in an area no larger than 2in x 2in.
  The tip will be placed in contact with the skin, and parameters may be adjusted throughout the treatment and will determined by the Clinician.

SUMMARY:
The intended use of the radiofrequency and microneedling devices used in this study is to assess the efficacy and safety of paired treatment for the treatment of facial aging.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are a healthy male or female 40 - 65 years of age. Up to 35 subjects will be enrolled at 2 study centers. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 4 treatments on the face.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 40 - 65 years old.
* Diagnosed with clinically evident moderate wrinkles and/or moderate photoaging, including but not limited to dyschromia, and willing to undergo treatments with the study devices.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* The subject is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is hypersensitive to light in the near infrared wavelength region.
* The subject is taking medication which is known to increase sensitivity to sunlight.
* The subject has a seizure disorders triggered by light.
* The subject is taking or have taken oral isotretinoin, such as Accutane®, within the last six months.
* The subject has an active localized or systemic infection, or an open wound in area being treated.
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated.
* The subject has active herpes simplex in the area being treated.
* The subject is receiving or have received gold therapy.
* The subject has a pacemaker.
* The subject has a metal implant that interferes with the transmission of energy to the electrical field.
* The subject has any embedded electronic devices that give or receive a signal such as Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant.
* The subject is allergic to adhesives such as glues on medical tape.
* The subject is allergic to gold.
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area or a neuropathic disorder.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated
* The subject is taking aspirin or are currently taking antiplatelets, thrombolytics, anti-inflammatories or anticoagulants.
* The subject has a history of bleeding coagulopathies.
* The subject is allergic to topical anesthetic.
* The subject has any of the following conditions:

  * Uncontrolled diabetes
  * Epilepsy
  * Autoimmune disease
  * HIV
  * Uncontrolled hypertension
* The subject has keloid formation propensity.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

* The subject has had unprotected sun exposure within four weeks of treatment, including the use of tanning beds or tanning products, such as creams, lotions, and sprays.
* The subject has a history of immunosuppression/immune deficiency or an auto-immune disorder.
* The subject is taking medications that alter the wound-healing response or evidence of compromised wound healing.
* The subject has a history of skin cancer or suspicious lesions in the treatment area.
* The subject has used retinoids in the last seven days in the area to be treated.
* The subject has used any chemical peels in the last three months in the treatment area.
* The subject has tattoos, permanent makeup, and permanent brows in the treatment area.
* The subject has received fillers or neurotoxin injections in the last two weeks.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Percent of Photos Identified Correctly of 30 Day Follow Up vs. Baseline | 30 day follow up
  The percent of correctly identified photographs (when comparing baseline photos vs. 30 day follow up photos) will be reported.
Percent of Photos Identified Correctly of 90 Day Follow Up vs. Baseline | 90 day follow up
  The percent of correctly identified photographs (when comparing baseline photos vs. 90 day follow up photos) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Director of Clinical Development
Locations (3):
- United States (3):
  - Center for Dermatology and Laser Surgery, Sacramento, California
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Laser & Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No